CLINICAL TRIAL: NCT01021657
Title: Lipid Profile of Tenon's Capsule in Glaucoma Patients
Brief Title: Lipid Profile of Tenon's Capsule
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Professor Catherine Creuzot-Garcher, Ophthalmology Department
Other Study IDs: Alain01
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2009-11-30 (Estimated); Status verified 2009-11

CONDITIONS: Glaucoma
Keywords: Glaucoma; Tenon's Capsule; Lipid profile; Assessment of lipid profile in Tenon's capsule in patients with Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Eye Tenon's Capsule
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glaucoma
  Interventions: Procedure: trabeculectomies, non penetrating deep sclerectomies

INTERVENTIONS:
Procedure: trabeculectomies, non penetrating deep sclerectomies

SUMMARY:
The purpose of this study is to provide data on the lipid profile of the Tenon's capsule in Human glaucomatous eyes and to establish possible relationships with the short term outcome of filtration surgery.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma
* Eligibility for surgery

Exclusion Criteria:

* Patients without Glaucoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient suffering from Glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To provide data on the lipid profile of the Tenon's capsule in Human glaucomatous eyes and to establish possible relationships with the short term outcome of filtration surgery. | 6 month later

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Creuzot-Gracher, MD, PhD, Principal Investigator — Ophthalmology unit CHU Dijon
Locations (1):
- Ophthalmology Unit CHU Dijon, Dijon, France